CLINICAL TRIAL: NCT03675529
Title: The Effect of Exercise on Tumor Hypoxia in Men With Localized Prostate Cancer Undergoing Radical Prostatectomy - a Randomized Controlled Pilot Study
Brief Title: The Effect of Exercise on Tumor Hypoxia in Men With Localized Prostate Cancer Undergoing Radical Prostatectomy.
Acronym: SHOR-TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sissal Sigmundsdóttir Djurhuus, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-18020711
Record Dates: First submitted 2018-08-24; First posted 2018-09-18 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: prostate neoplasm; exercise; high intensity interval training; tumor hypoxia; immune cells
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training bout (Experimental): Patients randomized to this group will perform a wattmax test immediately followed by 4 intervals of high and low intensity based on percentage of wattmax. Immediately after the exercise bout is finished patients will receive one dose of pimonidazole hydrochloride (500 mg per m2 body surface) in order to quantify tumor hypoxia by pathological analyses after removal of the prostate by radical prostatectomy the following day.
  Interventions: Behavioral: High Intensity Interval Training bout
- Controls (usual care) (No Intervention): Patients randomized to the control group will not be doing any exercise, but will after approximately 35 min from baseline blood sampling receive one dose of pimonidazole hydrochloride (500 mg per m2 bodysurface) in order to quantify tumor hypoxia by pathological analyses after removal of the prostate by radical prostatectomy the following day.

INTERVENTIONS:
Behavioral: High Intensity Interval Training bout — Patients randomized to the HIIT bout will perform one single supervised High Intensity Interval Training bout consisting firstly of a wattmax test on a stationary bike, in order to set the training intensity. This is followed by 10 minutes at low intensity at approximately 30% of wattmax. Subsequently patients will perform 16 min with 4 cycles with High and Low intensity. HI intervals consisting of 1 min with 100% of wattmax followed by 3 min recovery with the intensity load of 30% of wattmax.
  Arms: High Intensity Interval Training bout

SUMMARY:
Background and purpose: The purpose of this study is to investigate the effect of one acute exercise bout on tumor hypoxia in patients with localized prostate cancer undergoing radical prostatectomy.

The primary hypothesis is that exercise reduces tumor hypoxia and that the reduction is greater in patients performing one acute high intensity exercise bout compared to no training controls.

The investigators have not been able to identify any prior or current randomized trials investigating exercise and tumor hypoxia, and believe that such research is warranted and would be of great importance. Moreover there is a need for studies including biological measurements to allow a full assessment of the effect of exercise on diverse biomarkers and mechanistic pathways, which may influence cancer survival.

Subjects: Patients with histologically verified prostate adenocarcinoma scheduled for radical prostatectomy at Urologic Department, Rigshospitalet, Copenhagen, Denmark.

Methods: In this randomized controlled pilot study 30 patients with localized prostate cancer undergoing radical prostatectomy will be included and randomized 2:1 to either one single acute High Intensity Interval Training bout or usual care and no training the day prior to radical prostatectomy.

All patients will undergo assessment at inclusion (baseline) and the day prior to surgery.

Assessment includes: anthropometrics; blood pressure; resting hearth rate; hip and waist circumference, ECG, quality of life by self-report questionnaires; fasting blood sample measuring PSA (prostate specific antigen), cholesterol, triglycerides, insulin, c-peptide, HbA1c, glucose and inflammatory markers.

All patients will receive one dose of pimonidazole hydrochloride (500 mg per m2 body surface) in order to quantify tumor hypoxia by pathological analyses after removal of the prostate.

Biological tissue from tumor (primary prostate biopsies) will also be retrieved from the respective local pathological departments and from the perioperative prostate specimen and sent to protocol analyses.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of one acute exercise bout on tumor hypoxia in patients with localized prostate cancer randomized to one single acute I) High Intensity Interval Training bout compared to (II) usual care and no training prior to radical prostatectomy.

In addition to this the aim is to investigate the effect of one exercise bout on tumor vessel morphology and to investigate the effect of one acute exercise bout on intratumoral immune cell infiltration and to investigate the modulation of tumor-metabolism, -biology and signaling in patients randomized to either one acute High Intensity Interval Training bout compared to usual care and no training, the day prior to surgery.

Moreover this study will explore the acute response in immune cells, hormones and cytokines in blood samples taken before, during and after a single exercise session, and will collect physiological (metabolic profile and metabolic inflammatory markers) and psycho-social (e.g. fatigue, emotional well-being, anxiety) information regarding patients randomized to either one acute High Intensity Interval Training bout compared to usual care and no training, the day prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men with histologically verified localized prostate adenocarcinoma undergoing curative intended radical prostatectomy.

Exclusion Criteria:

* Age: <18 years
* Any other known malignancy requiring active treatment
* Performance status > 1
* Allergy to pimonidazole
* Ongoing treatment with beta blockers
* Physical disabilities precluding physical testing and/or exercise
* Inability to read and understand Danish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Tumor hypoxia | At prostatectomy
  Quantification of tumor hypoxia will be assessed using pimonidazole staining

SECONDARY OUTCOMES:
Intratumoral immune cell infiltration | Primary prostate biopsies and until radical prostatectomy
  Intratumoral immune cell infiltration will be quantified using histological analyses
Tumor vessel morphology | Primary prostate biopsies and until radical prostatectomy
  Tumor vessel morphology will be evaluated using histological analyses
Tumor metabolism-, biology and signaling | Primary prostate biopsies and until radical prostatectomy
  Tumor samples will undergo proteomic analyses in order to uncover potential upregulated biomarkers
Changes in immune cells during an acute exercise bout | From start of exercise bout and until 60 minutes post exercise
  Changes in immune cells during an acute exercise bout will be measured in blood samples using flowcytometry
Changes in epinephrine concentration | From start of exercise bout and until 60 minutes post exercise
  Concentration of epinephrine will be measured in blood samples by radioimmunoassay analyses.
Changes in nor-epinephrine concentration | From start of exercise bout and until 60 minutes post exercise
  Concentration of nor-epinephrine will be measured in blood samples by radioimmunoassay analyses.
Changes in various interleukines | From start of exercise bout and until 60 minutes post exercise
  Concentration of various interleukines will be measured in blood samples by measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in Tumor Necrosis Factor alpha (TNFa) concentration | From start of exercise bout and until 60 minutes post exercise
  Concentrations of TNFa will be measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in Interferon Gamma (IFNγ) concentration | From start of exercise bout and until 60 minutes post exercise
  Concentrations of IFNγ will be measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Concentration of C-reactive Protein (CRP) | Blood sampling on the day of radical prostatectomy
  Concentration of CRP will be measured in fasting blood sample by standard laboratory methods.
Total plasma cholesterol concentration | Blood sampling on the day of radical prostatectomy
  Concentrations of total cholesterol will be measured in fasting blood samples by standard laboratory methods.
Plasma LDL-Cholesterol concentration | Blood sampling on the day of radical prostatectomy
  Concentrations of LDL- cholesterol will be measured in fasting blood samples by standard laboratory methods.
Plasma HDL-Cholesterol concentration | Blood sampling on the day of radical prostatectomy
  Concentrations of HDL- cholesterol will be measured in fasting blood samples by standard laboratory methods.
Plasma triglyceride concentrations | Blood sampling on the day of radical prostatectomy
  Concentrations of triglycerides will be measured in fasting blood samples by standard laboratory methods.
HbA1C concentration | Blood sampling on the day of radical prostatectomy
  Concentrations of HbA1C will be measured in fasting blood samples by standard laboratory methods.
Plasma Insulin concentration | Blood sampling on the day of radical prostatectomy
  Concentrations of insulin will be measured in fasting blood samples by standard laboratory methods.
Plasma Glucose concentration | Blood sampling on the day of radical prostatectomy
  Concentrations of glucose will be measured in fasting blood samples by standard laboratory methods.
Wattmax-test | At baseline assessment
  The participants in the HIIT group will undergo a maximal graded exercise test on a bicycle ergometer for evaluation of cardiovascular function and determination of the maximum watt (wattmax). The test starts with a 3 min warm up at 70 watt (the watts may have to be adjusted to the individual fitness level). Warm up is immediately followed by a 20 watt increase every 1 min until exhaustion. The maximum watt will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sissal S Djurhuus, MD, Principal Investigator — PhD student
Locations (1):
- Center for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Djurhuus SS, Schauer T, Simonsen C, Toft BG, Jensen ARD, Erler JT, Roder MA, Hojman P, Brasso K, Christensen JF. Effects of acute exercise training on tumor outcomes in men with localized prostate cancer: A randomized controlled trial. Physiol Rep. 2022 Oct;10(19):e15408. doi: 10.14814/phy2.15408. PMID 36199257
- [Derived] Schauer T, Djurhuus SS, Simonsen C, Brasso K, Christensen JF. The effects of acute exercise and inflammation on immune function in early-stage prostate cancer. Brain Behav Immun Health. 2022 Sep 7;25:100508. doi: 10.1016/j.bbih.2022.100508. eCollection 2022 Nov. PMID 36133956